CLINICAL TRIAL: NCT05054673
Title: Clinical Performance of Newly Introduced Self-cured Universal Adhesive for Restoring Cervical Lesions in Geriatric Patients Over One Year (A Randomized Clinical Trial)
Brief Title: Clinical Performance of Self-cured Universal Adhesive for Restoring Cervical Lesions in Geriatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maysaa Mahmoud Mostafa Saad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: palfique bond
Record Dates: First submitted 2021-09-11; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Universal Adhesive

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): PALFIQUE universal adhesive (Tokuyama self-cure universal adhesive)
  Interventions: Other: universal adhesive
- control (Active Comparator): 3M™ ESPE™ single bond Universal Adhesive
  Interventions: Other: universal adhesive

INTERVENTIONS:
Other: universal adhesive — PALFIQUE universal adhesive
  Arms: intervention
Other: universal adhesive — 3M™ ESPE™ single bond Universal Adhesive
  Arms: control

SUMMARY:
the study is conducted to evaluate the clinical performance of PALFIQUE universal adhesive (Tokuyama self-cure universal adhesive), Versus 3m ESPE™ single bond Universal Adhesive, for restoring cervical lesions in geriatric patients over one year.

ELIGIBILITY:
Inclusion Criteria:

* The patient had to be in good general health
* Geriatric patients
* Have an acceptable oral hygiene level
* Class V cavities in anterior and posterior teeth
* Males & females included
* Anticipated availability for recalls (6 months and 12 months) through the 1-year study period

Exclusion Criteria:

* Lack of written informed consent to participate
* Poor oral hygiene,
* Severe bruxism
* Severe or chronic periodontitis
* Allergies to components of the materials used
* Underage patients
* Non vital pulp

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Measuring the Marginal adaptation | 1 year
  modified USPHS criteria, ordinal

SECONDARY OUTCOMES:
level of Retention | 1 year
  binary , modified USPHS criteria
Level of Marginal discoloration | 1 year
  ordinal, modified USPHS criteria
Rate of Secondary caries | 1 year
  binary , modified USPHS criteria
level of Postoperative sensitivity | 1 year
  binary , modified USPHS criteria